CLINICAL TRIAL: NCT04387357
Title: Multimodal Imaging in Alzheimer's Disease and Other Neurodegenerative Diseases
Brief Title: Multimodal Imaging in the Study of Disorientation in the Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Rostock (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Stefan Teipel, Prof. Dr. med, University Medical Center Rostock
Organization: University of Rostock (Other)
Other Study IDs: A-2012-0083
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Mild Cognitive Impairment; Dementia; Disorientation; Older Adults; Magnetic Resonance Imaging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Confusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Neurologically healthy older adults above the age of 50
- Experimental: Older adults above the age of 50 with Mild Cognitive Impairment or Dementia

SUMMARY:
The purpose of this study is to investigate whether markers of brain structure and function from MRI are associated with different levels of spatial orientation and gait parameters in people with mild cognitive impairment or dementia due to Alzheimer's disease when walking through a real world environment.

DETAILED DESCRIPTION:
This is an experimental cross-sectional study which primarily aims at identifying characteristic features of spatial disorientation among people with mild cognitive impairment and dementia. The features of interest are motion and physiological related changes that occur during instances of spatial disorientation, which will be derived from wearable sensors.

Additionally, brain structure and functional connectivity changes associated with different levels of spatial orientation and gait parameters will also be investigated through resting-state functional imaging.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and above
* Mini mental state examination (MMSE) ≥ 12 < 28 points for experimental group
* Mini mental state examination (MMSE) ≥ 28 points for control group
* Sufficient knowledge of German to understand participant information, declaration of consent and questionnaires
* Dated and signed declaration of consent
* Sufficient mobility and motivation to participate in the study

Exclusion Criteria:

* Less than 50 years
* Significantly impaired vision or hearing
* Severely reduced mobility: cannot move around independently (even with aids)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults and older adults with mild cognitive impairment or dementia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Spatial disorientation | Up to 3 years from start of the study
  Incidences of disorientation will be annotated in real-time using a customized annotation scheme in the pocket observer software

SECONDARY OUTCOMES:
Heart rate variability | Up to 3 years from start of the study
  Rate of change in heart rate will be measured using a wearable Photoplethysmography sensor
Skin conductance | Up to 3 years from start of the study
  Rate of change in electrodermal response will be measured using a wearable electrodermal activity sensor
Accelerometry | Up to 3 years from start of the study
  Incidences of change in movement behaviour and activity level will be measured using accelerometers
Grey matter volume | Up to 3 years from start of the study
  Rate of change in brain structural volume will be measured using a 3-Tesla scanner
White matter integrity | Up to 3 years from start of the study
  Rate of change in structural connectivity of brain white matter will be measured using a 3-Tesla scanner
Resting-state functional connectivity | Up to 3 years from start of the study
  Rate of change in functional connectivity of resting-state brain networks will be measured using a 3-Tesla scanner
Interview responses | Up to 3 years from start of the study
  Participants assessments of their sense of orientation are obtained using a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J. Teipel, Prof. Dr., Principal Investigator — University Medical Center Rostock
Locations (1):
- Clinic and Polyclinic for Psychosomatics and Psychotherapeutic Medicine, University Medical Center Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Schaat S, Koldrack P, Yordanova K, Kirste T, Teipel S. Real-Time Detection of Spatial Disorientation in Persons with Mild Cognitive Impairment and Dementia. Gerontology. 2020;66(1):85-94. doi: 10.1159/000500971. Epub 2019 Jul 30. PMID 31362286
- [Background] Ranasinghe KG, Hinkley LB, Beagle AJ, Mizuiri D, Dowling AF, Honma SM, Finucane MM, Scherling C, Miller BL, Nagarajan SS, Vossel KA. Regional functional connectivity predicts distinct cognitive impairments in Alzheimer's disease spectrum. Neuroimage Clin. 2014 Jul 23;5:385-95. doi: 10.1016/j.nicl.2014.07.006. eCollection 2014. PMID 25180158